CLINICAL TRIAL: NCT03829514
Title: Fenofibrate in Type 2 Diabetes- Novel Biomarkers and Mechanisms
Brief Title: Fenofibrate in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Timothy Lyons, Professor and Chief, Division of Endocrinology, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00079289
Record Dates: First submitted 2019-01-25; First posted 2019-02-04 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fenofibrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fenofibrate (Experimental): Single arm. Participants will take study medication
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — 40 patients (20 males and 20 females) aged 18-70 years, with type 2 diabetes and triglycerides >150 mg/dL will be recruited. They will have a physical exam and blood draw at visit 1. Participants will receive 160 mg fenofibrate to be taken orally daily for six weeks. They will return for a second visit after 6 weeks and have blood draw as follow up.
  Other Names: Trilipix; Triglide; Antara

SUMMARY:
Diabetic complications affecting the eyes, kidneys, and nerves are difficult to arrest once in progress. Recent evidence that fenofibrate confers a robust yet unexpected benefit in diabetic retinopathy offers an important translational research opportunity. The investigator's global proteomic study will provide new clues as to how fenofibrate protects vulnerable tissues, and will spur discovery of targets for new therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes of at least one year's duration; stable glycemic control (no more than 1.0% change in HbA1c in the previous six months, but no limit on HbA1c)
* Triglycerides >150 mg/dL (in the previous six months)

Exclusion Criteria:

* Previous use of Fenofibrate or other fibrates
* Pregnancy
* Active malignancy
* Recent cardiac event or congestive heart failure
* Active liver disease
* Significant renal impairment (serum creatinine > 2mg/dl)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fenofibrate
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fenofibrate
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Number of proteins and their relative abundance [Number; unit: proteins] | 667

OUTCOME MEASURES:

1. Primary Outcome: Number of Individual Plasma Proteins That Changed From Baseline to End-point Based on Limma T-Test of Protein Abundance as Determined by Proteomic Analysis Via Liquid Chromatography-mass Spectrometry
Description: Protein exclusive intensity values (counts/second) were normalized using cyclic loess normalization. Mean protein abundance as determined by the intensity for each protein was determined. 95% confidence intervals were calculated as a measure of dispersion. Paired means were compared using a Limma T-test and the p-value was adjusted for multiple comparisons using the Benjamini-Hochberg method. Mean Log2 Fold Change was calculated for each protein compared between 6 weeks and baseline. The number of proteins that changed between 6 weeks and baseline was zero.
Time Frame: Six weeks, from baseline visit to study completion visit
Population: One participant sample lacked quantity to test.
Measure: Mean (95% Confidence Interval); unit: Proteins
Units Other Than Participants: proteins
Arm/Group | Fenofibrate
Number analyzed (Participants) | 9
Number analyzed (proteins) | 667
Proteins | 0 [-2 to 2]
Statistical Analysis 1: Comparison: Fenofibrate; Test type: Other; p = 0.05, t-test, 2 sided; Signal intensity data were loess normalized and normalized data were used to perform a limma t-test with empirical Bayes smoothing to standard errors; Proteins were identified and quantified using EncyclopeDIA and visualized with Scaffold DIA using 1% false discovery thresholds at both the protein and peptide level. Protein exclusive intensity values were assessed for quality using an in-house ProteiNorm app, a tool for systematic evaluation of normalization methods, imputation of missing values and comparisons of multiple differential abundance methods . Cyclic loess normalization. The normalized data were used to perform statistical analysis using linear models for microarray data (limma) with empirical Bayes (eBayes) smoothing to the standard errors. Proteins with p-value < 0.05 were considered significant

ADVERSE EVENTS:
Time Frame: time each participate was receiving intervention; baseline and study completion, 6 weeks
Arm/Group | Fenofibrate
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT03829514/Prot_001.pdf
  • Informed Consent Form (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT03829514/ICF_002.pdf